CLINICAL TRIAL: NCT02672787
Title: A Randomized, ED-based Intervention to Improve Antihypertensive Adherence
Brief Title: A ED-based Intervention to Improve Antihypertensive Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Candace McNaughton, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 151384; K23HL125670 (NIH)
Record Dates: First submitted 2016-01-27; First posted 2016-02-03 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Hypertensive Emergency; Hypertension; Blood Pressure
Keywords: Antihypertensive adherence; Emergency medicine; Antihypertensives
MeSH Terms: conditions — Hypertensive Crisis; Hypertension | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ED usual care plus education (Active Comparator): ED usual care plus education
  Interventions: Behavioral: ED usual care plus education
- Intervention (Experimental): Subjects will receive the ED-based behavioral intervention
  Interventions: Behavioral: ED-based behavioral intervention

INTERVENTIONS:
Behavioral: ED-based behavioral intervention — Data collection, antihypertensive adherence assay, antihypertensive interview and EHR review, barrier identification, personalized goal setting, communication with PCP, and reminder messages/engagement messages.
  Arms: Intervention
Behavioral: ED usual care plus education — Data collection, antihypertensive adherence assay, antihypertensive interview, EHR review, and usual care education.
  Arms: ED usual care plus education

SUMMARY:
Despite great strides, hypertension remains an incredibly important disease and public health problem. This study addresses this critical need among ED patients, a unique population of patients who are (a) likely to benefit from an antihypertensive adherence intervention due to their high prevalence of uncontrolled blood pressure and poor adherence, and (b) at high risk for poor cardiovascular outcomes. The protocol provides for a multicomponent intervention bundle to be tested among ED patients. Successful clinic-based behavioral interventions generally target a combination of barriers to adherence; bundled interventions have shown success in a wide range of settings and diseases. In some cases, bundled components were necessary to achieve blood pressure benefit in a primary care setting; isolated educational efforts have had mixed success in the ED.

DETAILED DESCRIPTION:
More than 37 million Americans have uncontrolled hypertension, with associated costs of $93.5 billion in 2010. Emergency department visits for hypertension rose 25% from 2006 to 2011. According to the Centers for Disease Control and Prevention, "improved hypertension control…require[s] an expanded effort and an increased focus on blood pressure from health-care systems, clinicians, and individuals."

ED visits among patients with uncontrolled blood pressure are often missed opportunities for the ED to serve as an additional healthcare touchpoint and opportunity to impact chronic disease control by complementing chronic care. The ED is a common access point into the healthcare system, with more than 120 million visits annually among 20% of Americans. ED visits specifically for hypertension are also common, with more than 5 million visits per year and rising rapidly as more newly insured and chronically ill patients seek ED care. Elevated blood pressure (BP) is noted in 15-25% of all ED visits and cannot be attributed solely to pain. An ED-based intervention places focus on patients who are at increased risk for poor clinical outcomes and who are likely to gain benefit from interventions.

Medication adherence, or taking medications as prescribed, is crucial for BP control. Until now, measuring antihypertensive adherence in the ED has been limited to self-report, which is influenced by recall and social desirability biases and lack of an established patient-provider relationship. As a result, little is known regarding factors related to antihypertensive adherence or optimal interventions to improve adherence among ED patients. This project utilizes a validated mass spectrometry plasma assay as a measure of antihypertensive adherence to overcome these limitations. This tool will be combined with a conceptual framework in order to test our understanding of how adherence relates to blood pressure control among ED patients. The conceptual framework is based on work by Krousel-Wood, Bosworth, Murray, and Gellad and is grounded in the Information-Motivation-Behavioral Skills model of health behavior change, Social Cognitive Theory, and successful clinic-based adherence interventions.

ELIGIBILITY:
Inclusion Criteria:

1. <6 hours since initial evaluation by a treating physician in the ED
2. Prescribed only antihypertensives detected by the mass spectrometry plasma assay
3. Prescribed at least 1 antihypertensive detected by the mass spectrometry plasma assay
4. Functioning peripheral IV, available left over (after clinical testing) blood, or willing to undergo venipuncture to obtain blood
5. Anticipated discharge from the ED, per ED attending
6. Elevated blood pressure in the ED, including triage systolic blood pressure of at least 140 mmHg or triage diastolic blood pressure of at least 90 mmHg, or 2 or more elevated BP measurements after triage (>=140/90 mmHg)
7. Able and willing to complete ~45 minutes of surveys, discussion in the ED as well as return for 2 follow up visits (i.e., no plans to move away or change medical providers in the next 6 months)
8. Willing to receive reminder messages via chosen method (e.g., text, phone call, or letter) for 45 days after enrollment
9. Has a healthcare provider who prescribes blood pressure medication, defined as having had a clinic visit within the past year
10. Age ≥21 years and <85 years

Exclusion Criteria:

1. Received vasoactive medication (including prescribed BP medications) in the ED prior to enrollment
2. Previously enrolled
3. End stage renal disease or on hemodialysis
4. Known pregnancy or anticipated pregnancy within 6 months
5. Sepsis, acute blood loss, acute alcohol withdrawal, or inability to tolerate medications in the 24 hours prior to arrival
6. Unable to provide informed consent (e.g., altered mental status, chronic dementia, prisoner, or inability to speak/understand English)
7. Enrolled in home health or other chronic care coordination management plan

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-02; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
1-month Blood Pressure | 1-month
  The primary outcome is change in Blood Pressure, measured by BPTru, one month after enrollment.

SECONDARY OUTCOMES:
1-month Change in Adherence Measured by Assay | 1-month
  Change in adherence as measured by the plasma assay.
1-month Change in Adherence Measured by Patient-report | 1-month
  Change in adherence as measured by patient-report.
3-month Change in Blood Pressure | 3-month
  3-month Change in Blood Pressure, measured by BPTru
3-month Change in Adherence Measured by Patient-report | 3-month
  BP and patient-reported adherence will evaluate longer-term impact of the intervention.
Proportion of patients with controlled BP | 1-month
  Compare the proportion of patients who achieve controlled BP at 1-month
Proportion of patients with controlled BP | 3-month
  Compare the proportion of patients who achieve controlled BP at 3-month

OTHER OUTCOMES:
Association of death with antihypertensive adherence measured by the blood mass spectrometry assay | 1 year, minimum
  Evaluate whether adherence (by assay) predicts mortality among patients enrolled in the study
Association of death with antihypertensive adherence measured by patient report | 1 year, minimum
  Evaluate whether adherence (by patient report) predicts mortality among patients enrolled in the study
Association of repeat ED visits with antihypertensive adherence measured by the blood mass spectrometry assay | 1 year, minimum
  Evaluate whether adherence (by assay) predicts repeat ED visits, in survival analysis
Association of hospitalization with antihypertensive adherence measured by the blood mass spectrometry assay | 1 year, minimum
  Evaluate whether adherence (by assay) predicts hospitalization, in survival analysis
Impact of the intervention on patient trust, measured by the Primary Care Assessment Survey (PCAS), at 3 months, by study arm | 3 months
  Evaluate whether the intervention was associated with change in the trajectory of patient trust over 3 months (longitudinal analysis)
Relationship between intervention vs. usual care plus education on the change in measured side effects of antihypertensives (TOMHS survey) at 3 months | 3 months
  Evaluate whether the intervention or improvement in adherence were associated with higher patient-reported side effects, measured by the TOMHS, at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Candace McNaughton, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Spieker AJ, Nelson LA, Rothman RL, Roumie CL, Kripalani S, Coco J, Fabbri D, Levy P, Collins SP, Wang T, Liu D, McNaughton CD. Feasibility and Short-Term Effects of a Multi-Component Emergency Department Blood Pressure Intervention: A Pilot Randomized Trial. J Am Heart Assoc. 2022 Mar;11(5):e024339. doi: 10.1161/JAHA.121.024339. Epub 2022 Feb 23. PMID 35195015
- [Derived] Nelson LA, Spieker AJ, Kripalani S, Rothman RL, Roumie CL, Coco J, Fabbri D, Levy P, Collins SP, McNaughton CD. User preferences for and engagement with text messages to support antihypertensive medication adherence: Findings from a pilot study evaluating an emergency department-based behavioral intervention. Patient Educ Couns. 2022 Jun;105(6):1606-1613. doi: 10.1016/j.pec.2021.10.011. Epub 2021 Oct 12. PMID 34690012